CLINICAL TRIAL: NCT03317210
Title: Treatment of Anemia of Chronic Disease With True Iron Deficiency in Pregnancy
Brief Title: Intravenous Treatment of Anemia in Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34130203
Record Dates: First submitted 2017-06-23; First posted 2017-10-23 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Ferric Oxide, Saccharated; Epoetin Alfa

STUDY DESIGN:
Intervention Model Description: According to hemoglobin level at the start of the therapy, the women were either treated with intravenous iron and rhEPO or with intravenous iron only twice weekly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- iron therapy with good response (Other): Patients with an Hb level between 9.0 and 9.9 g/dl received 200 mg iron sucrose intravenously twice weekly. The maximum total iron dose was 1,600 mg, therefore therapy was stopped if the maximal iron sucrose dose was administered, or target Hb > 10.5 g/dL was achieved.
  Interventions: Drug: iron sucrose (200 mg VENOFER®)
- iron therapy with poor response (Other): Patients with an Hb level between 9.0 and 9.9 g/dl received 200 mg iron sucrose intravenously twice weekly. If response to therapy with iron sucrose was poor (i.e. Hb increase <0.7 g/dl after 2 weeks), patients additionally received recombinant human erythropoietin (10,000 U EPREX®, Janssen-Cilag, Baar, Switzerland).
  Interventions: Drug: iron sucrose (200 mg VENOFER®); Drug: recombinant human erythropoietin (10,000 U EPREX®)
- iron therapy and erythropoietin (Other): Patients with an Hb between 8.0 and 8.9 g/dl received 200mg iron sucrose and recombinant human erythropoietin intravenously twice weekly.
  Interventions: Drug: iron sucrose (200 mg VENOFER®); Drug: recombinant human erythropoietin (10,000 U EPREX®)

INTERVENTIONS:
Drug: iron sucrose (200 mg VENOFER®) — According to hemoglobin level at the start of the therapy, the women were either treated with intravenous iron and rhEPO or with intravenous iron only twice weekly.
  Other Names: Venofer
Drug: recombinant human erythropoietin (10,000 U EPREX®) — According to hemoglobin level at the start of the therapy, the women were treated with rhEPO twice weekly.
  Other Names: Eprex
  Arms: iron therapy and erythropoietin; iron therapy with poor response

SUMMARY:
The investigators assess and compare the efficacy of anemia treatment in pregnant women with anemia of chronic disease with true iron deficiency and in women with iron deficiency anemia.

DETAILED DESCRIPTION:
Fifty anemic pregnant women with moderate anemia were prospectively observed and treated in the Anemia clinic at the Department of Obstetrics, University Hospital Zurich. All patients had singleton pregnancies. All pregnant women fulfilled criteria of moderate iron deficiency anemia defined as hemoglobin (Hb) between 8.0 and 9.9 g/dl and serum ferritin <15 μg/l. In all women, the analyses of a blood count, iron status, erythropoietin, cross reactive protein (CRP), folic acid and vitamin B12 were conducted. According to hemoglobin level at the start of the therapy, the women were either treated with intravenous iron and rhEPO or with intravenous iron only twice weekly. Patients with an Hb level between 9.0 and 9.9 g/dl (33 patients) received 200 mg iron sucrose (VENOFER®, Vifor Int., St. Gallen, Switzerland) intravenously twice weekly (group A). If response to therapy was poor (i.e. Hb increase <0.7 g/dl) after 2 weeks (13 patients), patients additionally received rhEPO (10,000 U EPREX®, Janssen-Cilag, Baar, Switzerland) (group B). This cut-off for adequate primary response the investigators choose on the basis of previous experience. Patients with an Hb between 8.0 and 8.9 g/dl (17 patients) received iron sucrose (Venofer) and rhEPO (Eprex) twice weekly from the start of therapy (group C).

Sufficient overall response to therapy (the difference of baseline hemoglobin and after therapy) was defined as Hb increase >1.0 g/dl. The maximum total iron dose was 1,600 mg, therefore therapy was stopped if the maximal iron sucrose dose was administered, or target Hb > 10.5 g/dL was achieved.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with hemoglobin between 8.0 and 9.9 g/dl and serum ferritin <15 μg/l

Exclusion Criteria:

* vitamin B12 deficiency anemia
* folic acid deficiency anemia
* hemoglobinopathy
* multiples
* liver disease
* kidney disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-09-01 (Actual); Primary Completion 2006-07-31 (Actual); Study Completion 2006-07-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of Treatment: hemoglobin increase after therapy | 4 weeks
  In all women, the analyses of a blood count, iron status, erythropoietin, cross reactive protein (CRP), folic acid and vitamin B12 were conducted.The hematological parameters were checked twice a week in the anemia clinic and iron status once a week.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Zimmermann, Prof., Study Director — University of Zurich

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT03317210/Prot_SAP_000.pdf